CLINICAL TRIAL: NCT00950885
Title: Efficacy of Melatonin Treatment in a Phase Advance Model of Transient Insomnia
Brief Title: Melatonin Treatment for Induced Transient Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Charles Andrew Czeisler, MD, PhD, Baldino Professor of Sleep Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1R01HL093279 (NIH)
Record Dates: First submitted 2009-07-22; First posted 2009-08-03 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Delayed Sleep Phase Disorder; Jet-lag; Shift-work Disorder
Keywords: sleep; alertness; performance; vigilance; circadian
MeSH Terms: conditions — Jet Lag Syndrome | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): placebo control group will receive 4 doses of identically-appearing capsules containing cellulose
  Interventions: Biological: Placebo
- Low dose melatonin (Experimental): 0.5 mg melatonin
  Interventions: Biological: Low Dose Melatonin
- High dose melatonin (Experimental): 3.0 mg melatonin
  Interventions: Biological: High Dose Melatonin

INTERVENTIONS:
Biological: Low Dose Melatonin — Melatonin and placebo will be delivered as capsules on 4 successive days. All groups will receive placebo on days 1-3. Placebo group will continue to receive placebo on days 4, while low dose group will receive 0.5mg melatonin on day 4 and high dose group will receive 3.0mg melatonin on day 4.
  Arms: Low dose melatonin
Biological: Placebo — Melatonin and placebo will be delivered as capsules on 4 successive days. All groups will receive placebo on days 1-3. Placebo group will continue to receive placebo on days 4, while low dose group will receive 0.5mg melatonin on day 4 and high dose group will receive 3.0mg melatonin on day 4.
  Arms: Placebo
Biological: High Dose Melatonin — Melatonin and placebo will be delivered as capsules on 4 successive days. All groups will receive placebo on days 1-3. Placebo group will continue to receive placebo on days 4, while low dose group will receive 0.5mg melatonin on day 4 and high dose group will receive 3.0mg melatonin on day 4.
  Arms: High dose melatonin

SUMMARY:
Melatonin supplements have been reported to be an effective treatment for circadian rhythm sleep disorders, including shift work dyssomnia, jet-lag, delayed sleep phase syndrome, and sleep disruption suffered by many blind individuals. However, the mechanism(s) by which melatonin affects the timing of sleep are not well-understood. The purpose of this study is to determine if melatonin improves sleep and performance on a schedule simulating eastward travel. This study will provide information regarding the mechanism of action of melatonin that will be critical for the use of melatonin as a treatment for circadian rhythm sleep disorders.

DETAILED DESCRIPTION:
This study uses a randomized, double-blind, placebo-controlled, parallel groups design. The independent variable will be melatonin treatment group (0.3 mg melatonin, 3.0 mg melatonin, or placebo). Day of treatment will be an independent variable in analysis of sleep, cortisol, performance and alertness data. The primary outcome variables will be sleep efficiency and the peak of the plasma cortisol rhythm. Subjective and objective measures of alertness and performance during wake time will also be assessed as part of an exploratory analysis. Safety of short-term melatonin treatment will be assessed. The experimental protocol is divided into 5 segments, the ambulatory baseline segment, the laboratory adaptation segment, the initial constant posture (CP, to assess circadian phase), the melatonin/placebo intervention before advanced scheduled sleep, and second CP to assess final circadian phase.

The experimental protocol is divided into 5 segments, the ambulatory baseline segment, the laboratory adaptation segment, the initial constant posture (CP) for circadian phase assessment, the melatonin/placebo intervention, and a final post-treatment CP for assessment of circadian phase.

The Ambulatory Baseline consists of at least 21 days, outside the laboratory. During this segment, wrist activity and light levels will be recorded using an ambulatory recording device (Actiwatch-L) while the subject goes about his/her normal routine. During this segment, the subject will maintain a regular, self-selected sleep-wake/light-dark schedule (8h in bed, 16h awake), and a sleep diary. The subject will also call in to our time-stamped sleep-wake call-in telephone system just prior to each bedtime and immediately after each wake time.

The Laboratory Adaptation begins upon admission to the laboratory (Day 1 on protocol schematic in Figure 13) and continues until Day 3. The subject will be scheduled to sleep and wake at his/her regular times (determined during the ambulatory baseline). This segment of the study is designed to allow the subject to adapt to the laboratory environment and to allow all subjects to experience a standardized lighting regime prior to initial circadian phase assessment. We believe another reason the baseline days are essential is because prior to study individual subjects will experience varying light exposure patterns and levels. The standardized lighting conditions during baseline days allow stabilization of the subjects' circadian phase and phase of entrainment, and also control immediate lighting history prior to the study interventions. Ambient lighting during waking on the baseline days will be provided by ceiling panels and will be of ordinary indoor level, and all lights will be turned off (darkness) during the scheduled sleep episodes (black boxes on double raster plot of protocol). For all scheduled sleep episodes, polysomnographic recording of sleep will be taken. Due to the nature of the study, the exact timing of the beginning and ending of each study will be based on the individual subject's habitual sleep-wake schedule. Beginning on Day 1 of the study, saliva samples will be taken hourly during waking, and blood samples will be collected twice hourly for baseline melatonin and cortisol phase/amplitude estimation. Subjective alertness assessments will be collected twice per waking hour, and neurobehavioral performance testing will be conducted every 2 waking hours.

The initial Constant Posture (CP) circadian phase estimation begins eight hours before habitual sleep time on Day 3 and continues for 22 h (shown in the cross-hatched bars in Figure 13). Throughout the CP, the subject will be restricted to a semi-recumbent position in bed in very dim indoor light (see Lighting Conditions section below for description) and will be fed equivalent hourly snacks. This segment of the study is designed to allow assessment of circadian phase by either eliminating factors known or suspected to obscure or mask circadian rhythms (changes in posture, activity, food intake, light level) or by distributing such factors across all circadian phases. The subject will be attended by a trained staff member to ensure wakefulness throughout the CP. Collection of plasma melatonin and cortisol, subjective alertness and neurobehavioral performance data will continue as in the Laboratory Adaptation Segment. After the CP is complete, the subject will be allowed to be ambulatory for another 6 hours before an 8-hour sleep episode. We chose to use CPs rather than a Constant Routine in order to avoid sleep deprivation, the recovery from which would obscure the results of the treatment conditions.

The melatonin/placebo intervention days follow the initial CP. On experimental Day 4-5, scheduled sleep will occur 5 hours before habitual bedtime. Melatonin or placebo will be administered 30 minutes before lights-out. Twelve hours after waking the following day (Day 5), the CP to asses final circadian phase will begin and continue for 22 hours. The final sleep episode will be scheduled from 18:00 to 02:00 h to ensure that post-treatment phase estimates are in no way compromised by change of sleep time. Subjects will be informed that they are likely to experience sleep disruption, impaired alertness and other symptoms of jetlag for up to several days after they are discharged from the laboratory. Four hours after the CP on Day 7, the subject will be discharged home.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking for at least 6 months;
* Healthy (no medical, psychiatric or sleep disorders);
* No clinically significant deviations from normal in medical history, vital signs, physical examination, blood chemistry and hematology, and ECG;
* Women of childbearing potential must agree to use an acceptable method of birth control, and must have a negative serum pregnancy test;
* Body mass index of > 18 or < 30 kg/m2;
* No drugs or medication likely to affect sleep or alertness, as determined by the investigators;

Exclusion Criteria:

* History of alcohol or substance abuse;
* Positive result on drugs of abuse screening;
* Current or past history of sleep disorders, including but not limited to obstructive sleep apnea, or any significant sleep complaint;
* Psychiatric disorder, including a history of depression or dysthymia (characterized by depressed mood on the majority of days for at least two years);
* Recent acute or chronic medical disorder, including but not limited to hepatic impairment and severe chronic obstructive pulmonary disease;
* History of intolerance or hypersensitivity to melatonin or melatonin agonists;
* Pregnancy or lactation;
* Shift work in the last 3 years;
* Transmeridian travel (2 or more time zones) in past 3 months;
* Any other scientific or medical reason, as determined by the PI, such as non-compliance with protocol or intolerance to inpatient study conditions.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Circadian phase | Through the last 5 days of the study
Sleep efficiency | During sleep throughout the 7 day study

SECONDARY OUTCOMES:
Neurobehavioral performance | During wake throughout the 7 day study

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Czeisler, Ph.D., M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Per the NIH Policy on Resource Sharing, we will make the datasets collected in this grant available following publication of the final study results. Such datasets will not contain identifying information per the regulations outlined in HIPAA, and written permission will be obtained from those requesting the datasets.